CLINICAL TRIAL: NCT04874194
Title: Phase Ib/II Study of Omacetaxine and Venetoclax for Patients With Relapsed/Refractory Acute Myeloid Leukemia or Myelodysplastic Syndrome Harboring Mutant RUNX1
Brief Title: Omacetaxine and Venetoclax for the Treatment of Relapsed or Refractory Acute Myeloid Leukemia or Myelodysplastic Syndrome Harboring Mutant RUNX1
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study terminated early because the company was longer providing the investigational product.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0890; NCI-2021-03341 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0890 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-05-01; First posted 2021-05-05 (Actual); Results first posted 2025-11-03 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Recurrent Acute Biphenotypic Leukemia; Recurrent Acute Myeloid Leukemia; Recurrent Myelodysplastic Syndrome; Refractory Acute Biphenotypic Leukemia; Refractory Acute Myeloid Leukemia; Refractory Myelodysplastic Syndrome
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Biphenotypic, Acute; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Homoharringtonine; Esters; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Ph 1 Arm A (AML) Dose 0 (Experimental): Participants receive omacetaxine SC BID on days 2-4, and venetoclax PO on days 1-10 . Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Omacetaxine Mepesuccinate; Drug: Venetoclax
- Ph 1 Arm B (MDS) Dose 0 (Experimental): Participants receive omacetaxine SC BID on days 2-4, and venetoclax PO on days 1-10 . Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Omacetaxine Mepesuccinate; Drug: Venetoclax
- Ph 1 Arm A (AML) Dose +1 (Experimental): Participants receive omacetaxine SC BID on days 2-4, and venetoclax PO on days 1-14. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Omacetaxine Mepesuccinate; Drug: Venetoclax
- Ph 1 Arm B (MDS) Dose + 1 (Experimental): Participants receive omacetaxine SC BID on days 2-4, and venetoclax PO on days 1-14. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Omacetaxine Mepesuccinate; Drug: Venetoclax
- Ph 2 Arm A (AML) Dose +1 (Experimental): Participants receive omacetaxine SC BID on days 2-4, and venetoclax PO on days 1-14. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Omacetaxine Mepesuccinate; Drug: Venetoclax
- Ph 2 Arm B (MDS) Dose + 1 (Experimental): Participants receive omacetaxine SC BID on days 2-4, and venetoclax PO on days 1-14. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Omacetaxine Mepesuccinate; Drug: Venetoclax

INTERVENTIONS:
Drug: Omacetaxine Mepesuccinate — Given SC
  Other Names: Ceflatonin; Cephalotaxine, 4-methyl 2-hydroxy-2-(4-hydroxy-4-methylpentyl)butanedioate (ester), [3(R)]- (9CI); CGX-635; HHT; homoharringtonine; Synribo
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase Ib/II trial best dose, possible benefits and/or side effects of omacetaxine and venetoclax in treating patients with acute myeloid leukemia or myelodysplastic syndrome that has come back (recurrent) or does not respond to treatment (refractory) and have a genetic change RUNX1. Drugs used in chemotherapy, such as omacetaxine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Venetoclax may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. Giving omacetaxine and venetoclax may help to control the disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability and recommended phase 2 dose (RP2D) of omacetaxine in combination with venetoclax for patients with relapsed/refractory acute myeloid leukemia or myelodysplastic syndrome harboring a RUNX1 mutation. (Phase 1b) II. To determine the efficacy of omacetaxine in combination with venetoclax for patients with relapsed/refractory acute myeloid leukemia or myelodysplastic syndrome harboring a RUNX1 mutation. (Phase II)

SECONDARY OBJECTIVES:

I. To determine duration of response (DOR), event-free survival (EFS), and overall survival (OS).

II. To evaluate occurrence of minimal residual disease (MRD) negative status by multiparameter flow cytometry and molecular evaluation.

OUTLINE: This is a phase I, dose de-escalation study followed by a phase II study.

Patients receive omacetaxine subcutaneously (SC) twice daily (BID) on days 2-3 or 2-4, and venetoclax orally (PO) on days 1-7, 1-10 or 1-14. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up within 30 days, then every 3 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of relapsed or refractory acute myeloid leukemia (AML) (or biphenotypic or bilineage leukemia including a myeloid component) or myelodysplastic syndrome
* For myelodysplastic syndrome (MDS) patients, patients must have no response, progression, or relapse following at least 4 cycles of azacytidine or decitabine; and/or intolerance defined as grade >= 3 drug-related toxicity precluding continued therapy
* Age >= 18 years
* Subjects must have documented RUNX1 gene mutation
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Creatinine < 2 unless related to the disease
* Direct bilirubin < 2x upper limit of normal (ULN) unless increase is due to Gilbert's disease or leukemic involvement
* Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) < 3x ULN unless considered due to leukemic involvement
* In the absence of rapidly proliferative disease, the interval from prior treatment to time of initiation will be at least 7 days for cytotoxic or non-cytotoxic (i.e. immunotherapy) agents. Oral hydroxyurea and/or cytarabine (up to 2 g/m^2) for patients with rapidly proliferative disease is allowed before the start of study therapy, as needed, for clinical benefit and after discussion with the principal investigator (PI)
* Male subjects must agree to refrain from unprotected sex and sperm donation from initial study drug administration until 90 days after the last dose of study drug
* Willing and able to provide informed consent

Exclusion Criteria:

* Patients with t(15;17) karyotypic abnormality or acute promyelocytic leukemia (French-American-British [FAB] class M3-AML)
* Patients with any concurrent uncontrolled clinically significant medical condition including active infection or psychiatric illness, which could place the patient at unacceptable risk of study treatment
* Patients with active graft-versus-host-disease (GVHD) status post stem cell transplant (patients without active GVHD on chronic suppressive immunosuppression and/or phototherapy for chronic skin GVHD are permitted after discussion with the PI)
* Patients with any severe gastrointestinal or metabolic condition which could interfere with the absorption of oral study medications
* Known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection or known human immunodeficiency virus (HIV) infection
* Subject has a white blood cell count > 25 x 10^9/L. (Note: Hydroxyurea is permitted to meet this criterion.)
* Nursing women, women of childbearing potential (WOCBP) with positive urine pregnancy test, or women of childbearing potential who are not willing to maintain adequate contraception

  * Appropriate highly effective method(s) of contraception include oral or injectable hormonal birth control, intrauterine device (IUD), and double barrier methods (for example a condom in combination with a spermicide)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2024-09-16 (Actual); Study Completion 2024-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Courtney DiNardo, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] DiNardo CD, Jen WY, Montalban-Bravo G, Wang X, Loghavi S, Lavu S, Short NJ, Chien K, Issa GC, Pemmaraju N, Yilmaz M, Andreeff M, Borthakur G, Kadia TM, Daver NG, Garcia-Manero G, Mill CP, Su X, Fiskus W, Bhalla KN. Omacetaxine and venetoclax in relapsed/refractory acute myeloid leukemia or myelodysplastic syndrome with mutant RUNX1. Blood Neoplasia. 2025 Jul 25;2(4):100145. doi: 10.1016/j.bneo.2025.100145. eCollection 2025 Nov. PMID 40979071
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ph 1 Arm A (AML) Dose 0 | Ph 1 Arm B (MDS) Dose 0 | Ph 1 Arm A (AML) Dose +1 | Ph 1 Arm B (MDS) Dose + 1 | Ph 2 Arm A (AML) Dose +1 | Ph 2 Arm B (MDS) Dose + 1
Started | 3 | 2 | 9 | 0 | 10 | 0
Completed | 3 | 2 | 9 | 0 | 10 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: study moved to the phase 2 portion, with 10 AML patients treated at the RP2D. Due to lack of efficacy during an interim analysis, the AML arm was closed. In the phase 1b portion of the MDS arm, 2 patients were treated before the study was closed by the sponsor.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ph 1 Arm A (AML) Dose 0 | Ph 1 Arm B (MDS) Dose 0 | Ph 1 Arm A (AML) Dose +1 | Ph 1 Arm B (MDS) Dose + 1 | Ph 2 Arm A (AML) Dose +1 | Ph 2 Arm B (MDS) Dose + 1 | Total
Number analyzed (Participants) | 3 | 2 | 9 | 0 | 10 | 0 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 |  | 0 |  | 0
  Between 18 and 65 years | 0 | 1 | 5 |  | 3 |  | 9
  >=65 years | 3 | 1 | 4 |  | 7 |  | 15
Age, Continuous [Median (Full Range); unit: years] | 72 [66 to 84] | 70 [65 to 75] | 65 [29 to 75] |  | 73 [60 to 79] |  | 72 [29 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 3 |  | 6 |  | 9
  Male | 3 | 2 | 6 |  | 4 |  | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 |  | 0 |  | 0
  Asian | 0 | 0 | 1 |  | 0 |  | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 |  | 0 |  | 0
  Black or African American | 1 | 0 | 1 |  | 1 |  | 3
  White | 2 | 2 | 7 |  | 9 |  | 20
  More than one race | 0 | 0 | 0 |  | 0 |  | 0
  Unknown or Not Reported | 0 | 0 | 0 |  | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 9 |  | 10 |  | 24

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase 2 Dose (RP2D) of Omacetaxine in Combination With Venetoclax
Description: The RP2D will be selected at the end of the Phase 1b portion based on safety data , in Arms A and B independently. Preliminary efficacy and PK data for each dose level may also be considered as appropriate.
Time Frame: Up to 30 days
Population: RP2D was only assessed in the phase 1 portion of the study. In the phase 1b portion of the MDS arm, 2 patients were treated at dose level 0 before the study was closed by the sponsor.
Measure: Number; unit: mg/m2
Groups:
- Ph 1 Arm A (AML) Dose 0, Arm B (MDS) Dose 0, Arm A (AML) Dose +1: Participants receive omacetaxine SC BID on days 2-4, and venetoclax PO on days 1-10 . Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Omacetaxine Mepesuccinate: Given SC
  Venetoclax: Given PO
Arm/Group | Ph 1 Arm A (AML) Dose 0, Arm B (MDS) Dose 0, Arm A (AML) Dose +1 | Ph 1 Arm B (MDS) Dose + 1
Number analyzed (Participants) | 14 | 0
mg/m2
  Omacetaxine (days 2-4) | 1.25 |
  Venetoclax (days 1-14) | 400 |

2. Primary Outcome: Number of Participant to Achieve Complete Remission
Description: Complete Remission for AML is defined as: Absolute neutrophil count > 10^3/UL, platelets . 10^5/UL, red cell transfusion independence, absence of extramedullary disease, and bone marrow with < 5% blasts. Complete Remission for MDS is defined as: Absolute neutrophil count > 10^3/UL, platelets . 10^5/UL, hemoglobin >11 g/dl, and bone marrow with < 5% blasts. Peripheral dysplasia will be noted.
Time Frame: At day 28, and 3 cycles.
Population: Of the 24 patients enrolled in the study, three were not evaluable for response. One participant in Ph 1 Arm A (AML) Dose 0 was not evaluable for response. Two participants in Ph 2 Arm A (AML) Dose +1 were not available for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Ph 1 Arm A (AML) Dose 0 | Ph 1 Arm B (MDS) Dose 0 | Ph 1 Arm A (AML) Dose +1 | Ph 1 Arm B (MDS) Dose + 1 | Ph 2 Arm A (AML) Dose +1 | Ph 2 Arm B (MDS) Dose + 1
Number analyzed (Participants) | 2 | 2 | 9 | 0 | 8 | 0
Participants | 0 | 2 | 0 |  | 0 |

3. Secondary Outcome: Event-free Survival (EFS)
Description: Time from date of treatment start until the date of failure or death from any cause.
Time Frame: Up to Two years, 8 months, 30 days
Population: Due to lack of efficacy during an interim analysis, the AML arm was closed. In the phase 1b portion of the MDS arm, 2 patients were treated before the study was closed by the sponsor.
Measure: Median (Full Range); unit: Months
Arm/Group | Ph 1 Arm A (AML) Dose 0 | Ph 1 Arm B (MDS) Dose 0 | Ph 1 Arm A (AML) Dose +1 | Ph 1 Arm B (MDS) Dose + 1 | Ph 2 Arm A (AML) Dose +1 | Ph 2 Arm B (MDS) Dose + 1
Number analyzed (Participants) | 3 | 2 | 9 | 0 | 10 | 0
Months | 1.1 [0.6 to 3.4] | 16.8 [9.3 to 24.3] | 1.0 [0.6 to 2.8] |  | 1.1 [0.8 to 3.2] |

4. Secondary Outcome: Overall Survival (OS)
Description: The Kaplan-Meier method will be used to estimate the probabilities. Log-rank tests will be used to compare among subgroups of patients in terms of OS.
Time Frame: Up to Two years, 8 months, 30 days
Population: Due to lack of efficacy during an interim analysis, the AML arm was closed. In the phase 1b portion of the MDS arm, 2 patients were treated before the study was closed by the sponsor. Survival will be presented by median survival, which is the time point at which the cumulative survival drops below 50%. If there is no median survival (not reached), it means the cumulative survival was more than 50%.
Measure: Median (Full Range); unit: Months
Arm/Group | Ph 1 Arm A (AML) Dose 0 | Ph 1 Arm B (MDS) Dose 0 | Ph 1 Arm A (AML) Dose +1 | Ph 1 Arm B (MDS) Dose + 1 | Ph 2 Arm A (AML) Dose +1 | Ph 2 Arm B (MDS) Dose + 1
Number analyzed (Participants) | 3 | 2 | 9 | 0 | 10 | 0
Months | 9.4 [0.6 to 13.7] | NA [NA to NA] — Insufficient number of participants with events | 4.0 [1.1 to 9.2] |  | 3.4 [1.0 to 14.3] |

5. Secondary Outcome: Duration of Response
Description: Response date to loss of response or last follow up.
Time Frame: Up to Two years, 8 months, 30 days
Population: as for outcome 3
Measure: Median (Full Range); unit: Month
Arm/Group | Ph 1 Arm A (AML) Dose 0 | Ph 1 Arm B (MDS) Dose 0 | Ph 1 Arm A (AML) Dose +1 | Ph 1 Arm B (MDS) Dose + 1 | Ph 2 Arm A (AML) Dose +1 | Ph 2 Arm B (MDS) Dose + 1
Number analyzed (Participants) | 2 | 2 | 9 | 0 | 10 | 0
Month | NA [NA to NA] — insufficient number of participants with events | 15.0 [7.3 to 23.3] | NA [NA to NA] — insufficient number of participants with events |  | NA [NA to NA] — insufficient number of participants with events |

ADVERSE EVENTS:
Time Frame: Up to Two years, 8 months, 30 days
Description: There were zero participants at risk for Serious Adverse Events, Other Adverse Events and All-Cause Mortality for Ph 1 ARM B (MDS) Dose +1 and Ph 2 ARM B (MDS) Dose +1 due to the study closing and zero participants being registered on those two arms.
Arm/Group | Ph 1 Arm A (AML) Dose 0 | Ph 1 Arm B (MDS) Dose 0 | Ph 1 Arm A (AML) Dose +1 | Ph 1 Arm B (MDS) Dose + 1 | Ph 2 Arm A (AML) Dose +1 | Ph 2 Arm B (MDS) Dose + 1
All-Cause Mortality (participants affected / at risk) | 1/3 | 0/2 | 1/9 | 0/0 | 2/10 | 0/0
Serious Adverse Events (participants affected / at risk) | 3/3 | 2/2 | 5/9 | 0/0 | 7/10 | 0/0
Other Adverse Events (participants affected / at risk) | 1/3 | 1/2 | 5/9 | 0/0 | 4/10 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ph 1 Arm A (AML) Dose 0 (N=3) | Ph 1 Arm B (MDS) Dose 0 (N=2) | Ph 1 Arm A (AML) Dose +1 (N=9) | Ph 1 Arm B (MDS) Dose + 1 (N=0) | Ph 2 Arm A (AML) Dose +1 (N=10) | Ph 2 Arm B (MDS) Dose + 1 (N=0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-neutropenic fever (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Right middle cerebellar peduncle and medullary lesion - (Brain Lesions) (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Slurred speech (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Altered mental status (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute hypoxic respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis of the right toe (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ph 1 Arm A (AML) Dose 0 (N=3) | Ph 1 Arm B (MDS) Dose 0 (N=2) | Ph 1 Arm A (AML) Dose +1 (N=9) | Ph 1 Arm B (MDS) Dose + 1 (N=0) | Ph 2 Arm A (AML) Dose +1 (N=10) | Ph 2 Arm B (MDS) Dose + 1 (N=0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, specify (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-07): https://cdn.clinicaltrials.gov/large-docs/94/NCT04874194/Prot_SAP_001.pdf
  • Informed Consent Form (2023-03-16): https://cdn.clinicaltrials.gov/large-docs/94/NCT04874194/ICF_000.pdf